CLINICAL TRIAL: NCT00402675
Title: Leipzig Immediate Versus Early and Late PercutaneouS Coronary Intervention triAl in NSTEMI - LIPSIA-NSTEMI TRIAL
Brief Title: Randomized Trial of Immediate Versus Early and Selective Invasive Percutaneous Coronary Intervention in NSTEMI
Acronym: LIPSIA-NSTEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Holger Thiele, University of Leipzig - Heart Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leipzig-4
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2006-11

CONDITIONS: Myocardial Infarction
Keywords: NSTEMI; infarction; treatment; percutaneous coronary intervention; non-ST-elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate Intervention (Active Comparator): Patients with NSTEMI undergo immediate invasive angiography (< 2 hours)
  Interventions: Procedure: Timing of percutaneous coronary intervention
- Early Intervention (Active Comparator): Patients with NSTEMI undergo early invasive angiography (12-48 hours)
  Interventions: Procedure: Timing of percutaneous coronary intervention
- Selective invasive angiography (Active Comparator): Patients with NSTEMI undergo selective invasive angiography
  Interventions: Procedure: Timing of percutaneous coronary intervention

INTERVENTIONS:
Procedure: Timing of percutaneous coronary intervention — Immediate, early or selective invasive angiography

SUMMARY:
In non-ST-elevation the optimal time of percutaneous coronary intervention (PCI) is unclear.

Some studies showed benefit of very early PCI, some others early PCI between 12-48 hours and others even showed a benefit of a selective invasive approach only in case of recurrence of symptoms or a positive stress test.

The optimal timing of intervention is still matter of debate as a result of a randomized clinical trial.

DETAILED DESCRIPTION:
In this randomized, controlled, open-label clinical trial we compare a very early cardiac catheterization (< 2,5 hours after randomization) similar to ST-elevation myocardial infarction treatment, versus an early invasive approach (within 2-48 hours after randomization) versus a selective invasive approach in patients with non-ST-elevation myocardial infarction.

All patients are treated with heparin, ASA, Clopidogrel loading dose (600 mg) with subsequent 75 mg/d and tirofiban for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms:

   Instable angina pectoris:
   * Angina at rest < 24 hours
   * new onset worsening angina within the last weeks with angina at very low threshold < 24 h
2. Troponin T:

   Troponin T-elevation ≥ 0,03 μg/l
3. Informed consent

Exclusion Criteria:

1. Age < 18 years
2. Age > 90 years
3. STEMI
4. Hemodynamic instability
5. Cardiogenic shock
6. Warfarin therapy
7. Contraindications for GpIIb/IIIa-inhibitors
8. life expectancy < 6 months
9. known high bleeding risk
10. Pregnancy
11. Other reasons for Troponin-elevation: Myocarditis, secondary after hypertensive crisis, cardiac decompensation
12. No informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
peak creatine kinase- MB level | 5 days

SECONDARY OUTCOMES:
Major bleeding complications (GUSTO definition) | 30 days
Composite: death, re-myocardial infarction, recurrent unstable angina | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (5):
- Germany (5):
  - Klinikum Links der Weser, Bremen
  - Städt. Klinikum St. Georg, Leipzig
  - University of Leipzig - Heart Center, Leipzig
  - University of Leipzig, Leipzig
  - Krankenhaus der Barmherzigen Brüder, Regensburg

REFERENCES:
- [Derived] Thiele H, Rach J, Klein N, Pfeiffer D, Hartmann A, Hambrecht R, Sick P, Eitel I, Desch S, Schuler G; LIPSIA-NSTEMI Trial Group. Optimal timing of invasive angiography in stable non-ST-elevation myocardial infarction: the Leipzig Immediate versus early and late PercutaneouS coronary Intervention triAl in NSTEMI (LIPSIA-NSTEMI Trial). Eur Heart J. 2012 Aug;33(16):2035-43. doi: 10.1093/eurheartj/ehr418. Epub 2011 Nov 21. PMID 22108830